CLINICAL TRIAL: NCT01949636
Title: An fMRI Test of the Dynamic Vulnerability Model of Obesity: Risk Factor Plasticity
Brief Title: The Chocolate Study
Status: Completed | Type: Observational
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 092468; R01DK092468 (NIH)
Record Dates: First submitted 2013-07-18; First posted 2013-09-24 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- lean adolescents
  Interventions: Other: Functional Magnetic Resonance Imaging

INTERVENTIONS:
Other: Functional Magnetic Resonance Imaging

SUMMARY:
The purpose of this study is to test the dynamic vulnerability model of obesity using brain imaging.

DETAILED DESCRIPTION:
Obese vs lean humans show greater gustatory/oral somatosensory and reward region responsivity to palatable food images/cues and this predicts future weight gain (Yokum et al., 2011; Stice et al., 2008, 2010b; Stoeckel et al., 2008), in line with reward surfeit and incentive sensitization models of obesity (Berridge, 2009; Davis et al., 2004). Yet, obese vs lean humans have fewer dopamine (DA) receptors in striatal reward regions, show reduced striatal response to palatable food intake, and low striatal response predicts future weight gain in those at genetic risk for reduced DA signaling (Felsted et al., 2010; Stice et al., 2008; Wang et al., 2001; Volkow et al., 2008), in line with the reward deficit model of obesity (Wang et al., 2002b). One explanation for the mixed findings is that some of these findings reflect initial risk factors and others result from overeating. Firing of DA neurons in reward regions shifts from food intake to cues that predict food intake after conditioning (Kiyatkin et al., 1994; Schultz et al., 1993) and overeating leads to reduced D2 receptor density, D2 sensitivity, and reward sensitivity in rats (Alsio et al., 2010; Kelley et al., 2003; Johnson & Kenny, 2010) and striatal response to food in humans (Stice et al., 2010a), implying that overeating leads to increased incentive sensitization and down-regulation of reward regions. Further, reduced inhibitory region response to food images/cues predicts future overeating and weight gain (Cornier et al., 2010). Data imply that youth at risk for obesity initially show greater responsivity of regions that encode the reward value of food cues, coupled with greater responsivity of gustatory/oral somatosensory regions that encode the sugar and fat content of foods, and with reduced inhibitory region responsivity, which lead to overeating/weight gain that produces blunted striatal DA signaling, increased responsivity of reward valuation regions to food cues, and reduced inhibitory activation in response to food stimuli, increasing risk for further overeating/weight gain. We propose to conduct a rigorous test of this dynamic-vulnerability model using a novel repeated measures fMRI design in which teens complete scans annually over 4 years. Aim 1: test whether elevated gustatory/oral somatosensory and reward region responsivity and reduced inhibitory region responsivity to palatable food images, cues, and intake of food varying in sugar/fat content, and behavioral inhibitory control deficits/immediate reward bias predict initial increases in % body fat in 130 lean teens. Aim 2: use growth curve models to test whether initial increases in % body fat and energy dense food intake predict future decreases in striatal response to palatable food receipt, increases in reward circuitry response to palatable food images/cues, decreased inhibitory region response to food images/cues, and increased behavioral inhibitory control deficits/immediate reward bias. Aim 3: test whether decreased striatal response to palatable food, increased reward region response to food images/cues, reduced inhibitory region response to food images/cues, behavioral inhibitory control deficits/immediate reward bias predict further escalation in % body fat.

ELIGIBILITY:
Inclusion Criteria:

* between 14-16 years old
* BMI between 25th and 75th percentile

Exclusion Criteria:

* contraindicators of functional magnetic resonance imaging (fMRI)

  1. metal implants
  2. braces
  3. pregnancy
* symptoms of major psychiatric disorders (substance use disorders, conduct disorder, attention deficit hyperactive disorder, major depression, bipolar disorder, panic disorder, agoraphobia, generalized anxiety disorder)
* binge eating
* use of pyschoactive drugs
* serious medical conditions (diabetes, brain injury)
* smoking
* dietary allergy to dairy

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 130 lean adolescents between 14-16 years old with BMIs between the 25th and 75th percentile at baseline
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2012-05; Primary Completion 2016-06 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
increases in BMI | 1, 2, 3, and 4 years
  Whether increases in BMI are predicted by: elevated reward region responsivity and reduced inhibitory region responsivity to palatable food varying in sugar/fat content (measured during fMRI scan)

SECONDARY OUTCOMES:
striatal response to palatable food receipt; reward response and inhibitory response to palatable food cues, and inhibitory control deficits/immediate reward bias | 1, 2, 3, and 4 years
  whether increases in BMI and food intake predict: decreased striatal response to palatable food receipt, increased reward response and decreased inhibitory response to palatable food cues, and increased inhibitory control deficits/immediate reward bias (as measured during fMRI scan assessment).

OTHER OUTCOMES:
increases in BMI | 4 years
  whether future increases in BMI (measured at 3 year follow-up) is predicted by: decreased striatal response to palatable food, increased reward response to food cues, reduced inhibitory response to food cues, and behavioral inhibitory control deficits/immediate reward bias (as measured in fMRI scan assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stice, Ph.D., Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Portland, Oregon, United States

REFERENCES:
- [Background] Alsio J, Olszewski PK, Norback AH, Gunnarsson ZE, Levine AS, Pickering C, Schioth HB. Dopamine D1 receptor gene expression decreases in the nucleus accumbens upon long-term exposure to palatable food and differs depending on diet-induced obesity phenotype in rats. Neuroscience. 2010 Dec 15;171(3):779-87. doi: 10.1016/j.neuroscience.2010.09.046. Epub 2010 Sep 26. PMID 20875839
- [Background] Berridge KC. 'Liking' and 'wanting' food rewards: brain substrates and roles in eating disorders. Physiol Behav. 2009 Jul 14;97(5):537-50. doi: 10.1016/j.physbeh.2009.02.044. Epub 2009 Mar 29. PMID 19336238
- [Background] Cornier MA, Salzberg AK, Endly DC, Bessesen DH, Tregellas JR. Sex-based differences in the behavioral and neuronal responses to food. Physiol Behav. 2010 Mar 30;99(4):538-43. doi: 10.1016/j.physbeh.2010.01.008. Epub 2010 Jan 22. PMID 20096712
- [Background] Davis C, Strachan S, Berkson M. Sensitivity to reward: implications for overeating and overweight. Appetite. 2004 Apr;42(2):131-8. doi: 10.1016/j.appet.2003.07.004. PMID 15010176
- [Background] Felsted JA, Ren X, Chouinard-Decorte F, Small DM. Genetically determined differences in brain response to a primary food reward. J Neurosci. 2010 Feb 17;30(7):2428-32. doi: 10.1523/JNEUROSCI.5483-09.2010. PMID 20164326
- [Background] Johnson PM, Kenny PJ. Dopamine D2 receptors in addiction-like reward dysfunction and compulsive eating in obese rats. Nat Neurosci. 2010 May;13(5):635-41. doi: 10.1038/nn.2519. Epub 2010 Mar 28. PMID 20348917
- [Background] Kelley AE, Will MJ, Steininger TL, Zhang M, Haber SN. Restricted daily consumption of a highly palatable food (chocolate Ensure(R)) alters striatal enkephalin gene expression. Eur J Neurosci. 2003 Nov;18(9):2592-8. doi: 10.1046/j.1460-9568.2003.02991.x. PMID 14622160
- [Background] Kiyatkin EA, Gratton A. Electrochemical monitoring of extracellular dopamine in nucleus accumbens of rats lever-pressing for food. Brain Res. 1994 Aug 1;652(2):225-34. doi: 10.1016/0006-8993(94)90231-3. PMID 7953734
- [Background] Schultz W, Apicella P, Ljungberg T. Responses of monkey dopamine neurons to reward and conditioned stimuli during successive steps of learning a delayed response task. J Neurosci. 1993 Mar;13(3):900-13. doi: 10.1523/JNEUROSCI.13-03-00900.1993. PMID 8441015
- [Background] Stice E, Davis K, Miller NP, Marti CN. Fasting increases risk for onset of binge eating and bulimic pathology: a 5-year prospective study. J Abnorm Psychol. 2008 Nov;117(4):941-6. doi: 10.1037/a0013644. PMID 19025239
- [Background] Stice E, Yokum S, Blum K, Bohon C. Weight gain is associated with reduced striatal response to palatable food. J Neurosci. 2010 Sep 29;30(39):13105-9. doi: 10.1523/JNEUROSCI.2105-10.2010. PMID 20881128
- [Background] Stice E, Yokum S, Bohon C, Marti N, Smolen A. Reward circuitry responsivity to food predicts future increases in body mass: moderating effects of DRD2 and DRD4. Neuroimage. 2010 May 1;50(4):1618-25. doi: 10.1016/j.neuroimage.2010.01.081. Epub 2010 Jan 29. PMID 20116437
- [Background] Stoeckel LE, Weller RE, Cook EW 3rd, Twieg DB, Knowlton RC, Cox JE. Widespread reward-system activation in obese women in response to pictures of high-calorie foods. Neuroimage. 2008 Jun;41(2):636-47. doi: 10.1016/j.neuroimage.2008.02.031. Epub 2008 Mar 4. PMID 18413289
- [Background] Volkow ND, Wang GJ, Telang F, Fowler JS, Thanos PK, Logan J, Alexoff D, Ding YS, Wong C, Ma Y, Pradhan K. Low dopamine striatal D2 receptors are associated with prefrontal metabolism in obese subjects: possible contributing factors. Neuroimage. 2008 Oct 1;42(4):1537-43. doi: 10.1016/j.neuroimage.2008.06.002. Epub 2008 Jun 13. PMID 18598772
- [Background] Wang GJ, Volkow ND, Felder C, Fowler JS, Levy AV, Pappas NR, Wong CT, Zhu W, Netusil N. Enhanced resting activity of the oral somatosensory cortex in obese subjects. Neuroreport. 2002 Jul 2;13(9):1151-5. doi: 10.1097/00001756-200207020-00016. PMID 12151759
- [Background] Wang GJ, Volkow ND, Logan J, Pappas NR, Wong CT, Zhu W, Netusil N, Fowler JS. Brain dopamine and obesity. Lancet. 2001 Feb 3;357(9253):354-7. doi: 10.1016/s0140-6736(00)03643-6. PMID 11210998
- [Background] Yokum S, Ng J, Stice E. Attentional bias to food images associated with elevated weight and future weight gain: an fMRI study. Obesity (Silver Spring). 2011 Sep;19(9):1775-83. doi: 10.1038/oby.2011.168. Epub 2011 Jun 16. PMID 21681221
- [Derived] Yokum S, Bohon C, Berkman E, Stice E. Test-retest reliability of functional MRI food receipt, anticipated receipt, and picture tasks. Am J Clin Nutr. 2021 Aug 2;114(2):764-779. doi: 10.1093/ajcn/nqab096. PMID 33851199
- [Derived] Yokum S, Stice E. Weight gain is associated with changes in neural response to palatable food tastes varying in sugar and fat and palatable food images: a repeated-measures fMRI study. Am J Clin Nutr. 2019 Dec 1;110(6):1275-1286. doi: 10.1093/ajcn/nqz204. PMID 31535135
- [Derived] Shearrer GE, Stice E, Burger KS. Adolescents at high risk of obesity show greater striatal response to increased sugar content in milkshakes. Am J Clin Nutr. 2018 Jun 1;107(6):859-866. doi: 10.1093/ajcn/nqy050. PMID 29771283
- See also: Recruitment website — http://chocolate.ori.org/